CLINICAL TRIAL: NCT03216200
Title: A Single Center Open Label Early Feasibility Study to Evaluate the Efficacy and Safety of the RenewalNail™ Plasma Treatment System in Patients With Mild to Moderate Onychomycosis (Fungal Nail) of the Hallux Caused by Trichophyton Rubrum or Trichophyton Mentagrophytes.
Brief Title: Early Feasibility Study to Evaluate the Efficacy of the RenewalNail™ Plasma Treatment System in Patients With Onychomycosis (Fungal Nail)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeviceFarm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFCR-0003
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Onychomycosis of Toenail; Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: single center open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): 5 Subjects with 20-75% Distal Subungual Onychomycosis (mild to moderate DSO) infection of their big toe (hallux) nail infected by the dermatophytes Trichophyton (T.) rubrum or T. mentagrophytes will be enrolled. All Subjects will receive three 45-minute plasma treatments performed over a week.
  Interventions: Device: plasma treatment

INTERVENTIONS:
Device: plasma treatment — application of cold atmospheric plasma to a fungal infected toenail
  Other Names: RenewalNail™ plasma treatment system

SUMMARY:
A study to determine if a three-treatment protocol with the RenewalNail™ plasma treatment system over a week will result in mycological cure and/or clear nail growth on the treated hallux toe.

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical feasibility of DeviceFarm, Inc.'s RenewalNail™ system and the treatment protocol that was developed based on extensive laboratory testing on human cadaver nails. The Protocol calls for three 45-minute treatments performed over a week to achieve mycological cure. Mycological cure will be assessed with two consecutive mycological culture tests done over a week following the third treatment. Two consecutive negative mycology culture results confirm the elimination of fungus causing onychomycosis infection, as recommended by recent FDA guidance. There will be no placebo arm in the study. Clear nail growth will be documented and assessed by photography for 5 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are between 21 to 75 years (inclusive) of age;
* Subjects who are in good general health and free from any clinically significant disease that might interfere with the study evaluations;
* Subjects with established clinical diagnosis of distal subungual onychomycosis;
* Subjects with at least one big toe nail involved with 20-75% infection;
* Subjects with both positive KOH and culture for onychomycosis dermatophytes in screening of nail samples;
* Subjects whose infection is confirmed to be caused by T. rubrum or T. mentagrophytes;
* Subjects who are willing and able to refrain from employing other (non-study) treatments (traditional or alternative) for his or her toenail onychomycosis throughout study participation;
* Subjects who are willing and able to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers during the week of treatment (from Study Visits 1 through 3);
* Subjects who are willing and able to give written informed consent and able to adhere to procedures and visit schedules;
* Women of childbearing potential who are currently sexually active must agree to use a medically accepted method of contraception while receiving protocol specified treatment. Methods include condoms (male or female), diaphragm or cervical cap with spermicide, medically prescribed intrauterine device, oral or systemic hormonal contraceptive, surgical sterilization (e.g., hysterectomy or tubal ligation);
* Women of childbearing potential who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study;
* Women of childbearing potential must have a negative pregnancy test prior to start of study.

Exclusion Criteria:

* Subjects with onychomycosis infection involving lunula of the affected toenail(s) or spikes of disease extending to nail matrix in the affected big toenail;
* Subjects whose foot is too large (larger than US men's size 13) or too small (smaller than US women's size 3) to properly fit into the plasma treatment device;
* Subjects whose affected big toenail cannot become normal in the opinion of the investigator;
* Subjects who received topical antifungal treatment of the nails within 2 weeks before study initiation;
* Subjects who received systemic antifungal treatment within 3 months before study initiation;
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding treatment;
* Subjects who are immunocompromised (e.g. adrenal insufficiency, diabetes mellitus, febrile neutropenia, and the human immunodeficiency virus infected);
* Subjects with any pacemakers, or any metallic implants or prostheses in the vicinity of the treatment site (such as ankle, foot, etc.);
* Subjects with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study;
* Subjects who feel they cannot sit for 45 minutes at a time during the treatment;
* Subjects who are part of the staff personnel directly involved with this study or who are family members of the investigational study staff;
* Subjects with known allergy to any of the tested treatment products [i.e. perfluorocarbons and plastic polycarbonate];
* Women who are pregnant, breastfeeding, or planning pregnancy prior to the end of study participation;

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N Roe, PhD, Principal Investigator — DeviceFarm, Inc.
Locations (1):
- David L. Kahan, DPM, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 54 [48 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Mycological Cure
Description: number of participants with mycological cure defined as two consecutive negative cultures per FDA guideline
Time Frame: 2 cultures taken a week apart within 2 weeks after the first treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Clear Nail Growth
Description: Number of patients with photographic evidence of increased clear nail growth
Time Frame: 5 months after the first treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 3

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03216200/Prot_000.pdf